CLINICAL TRIAL: NCT03254641
Title: Calciotropic Effects After HCG Stimulation Test
Status: Completed | Type: Observational
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, MD, group leader, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-17004362
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2020-10

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hypogondal men: men referred for hCG stimulation test
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — 5000 IE times one
  Other Names: hCG

SUMMARY:
We have in a pilot study found that serum calcium levels change in response to hCG stimulation test. We observed that serum calcium level measured at baseline and 72 hours after hCG stimulation were different in men with gonadal insufficiency referred for this stimulation test. Now we want to investigate a large cohort of men referred for hCG stimulation test due to suspected impaired gonadal function.

DETAILED DESCRIPTION:
Introduction:

hCG signals through the LHCGR receptor and is know to stimulate testosterone production. hCG stimulation tests are therefore used to evaulate the capacity of the testis to respond to LH/hCG and thereby determine the degree og gonadal insufficiency and need for testosterone supplementation. Some groups have found LHCRG in extragondal tissues indicating a direct effect of hCG/LH outside the gonads. We noticed that some men with gonadal insuffciency had a low calcium level after hCG stimulation test. Now we would like to investigate whether this putative effect on calcium homeostasis of hCG is due to a direct effect or an indirect effect through testosterone or other sex steroids that also change in response to hCG stimulation. Moreover, we would like to clarify whether the chnage in calcium is compensated by classical regulators such as PTH, 1,25OH2D3, calcitonin, phosphate, CTX, alkaline phosphatase or other factors.

Aim of study:

The purpose of this study is to describe changes in calcium and calciotropic hormones after hCG stimulation test

DESIGN This is a prospective observational study

Patients and methods 100 men referred for hCG stimulation test due to suspected gonadal insuffciency age 18-60 years at Department of growth and reproduction, Rigshospitalet

Exclusion criteria are

intake of high dose calcium (above 1 mg daily) Known Disorders related to calcium metabolism, hypercalcemia, Granulomatous disease such as Wegener, tuberculosis, etc,

SAMPLE SIZE CALCULATION AND STATISTICS By using a test level of 5% (level of significance), power of 80% and at least 100 men completing the trial will enable us to detect a change in calcium of 10%, and a change in serum PTH of 30%.

SCREENING AND TIME COURSE Men referred for hCG stimulation test at ourDepartment will be screened for eligibility to the study. Those who meet the criteria for participation will be informed, and if they consent allocated to the study.

Each person will have one blood sampling performed prior to the test and 72 and 96 hours after the test.

Blood samples Venus blood is drawn preoperatively before hCG administration, 72 and 96 hours after. Serum will be send for analysis within 45 minutes and the rest frozen within 1 hour and will be stored at minus 20 degrees celsius until analysis.

OUTCOME MEASUREMENTS

Primary endpoints

•Changes in total, albumin corrected and ionized calcium

Main Secondary endpoints

* Changes in PTH
* Changes in 1,25OH2D3
* Changes in Phosphate
* Changes in FGF23
* Changes in Calcitonin
* Changes in LHCGR in serum
* Changes in Cortisol
* Changes in total and free testosterone
* Changes in total and free estradiol
* Changes in kidney function (GFR/creatinin)
* Changes in gonadotropins
* Changes in 25OHD, 24,25OH2D3
* Changes in serum concentrations of putative regulators and downstream signals osteocalcin, osteopontin, RANKL, osteoprotegerin (OPG), alpha Klotho, Sclerostin and IGF-1.

Temporal changes in serum level of binding proteins. differences for vitamin D binding protein, albumin and sex hormone binding globulin.

Predefined subgroups orchiectomized men/ bilaterally irradiated testis High versus low baseline estradiol/testosterone Low/high calcium/PTH baseline

ANALYSIS AND INTERVENTION

Reproductive hormones and growth factors will be analysed at dept. of GR, Rigshospitalet. Other serum analyses will be analysed at Department of clinical biochemistry, and Aarhus Kommune Hospital

ETHICS AND SIDE EFFECTS All the patients will have full-filled their investigation, before they are invited to the study. They will be informed of potential adverse effects, and they can leave the trial at any point without any consequences. This study poses no additional risk to the patients except for the blood samples as everything else is according to standard clinical practice.

PUBLICATION OF RESULTS All results, positive or negative will be submitted to peer reviewed scientific journals. Data will successively be obtained and transferred to a statistical database.

ELIGIBILITY:
Inclusion Criteria:

- men aged 18-60 years referred for hCG stimulation test due to previous treatment for testis cancer

Exclusion Criteria:

* high intake calcium
* know disorders in calcium homeostasis

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — referred for hCG stimulation test
Study Population: men with suspected gonadal i suffciency ofter after orchiectomy or bilateral irradiation due to testis cancer
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
change in total, albumin corrected or ionized calcium | 72 and 96 hours after hCG injection
  mmol/l

SECONDARY OUTCOMES:
PTH | 72 and 96 hours after hCG injection
1,25OH2D3 | 72 and 96 hours after hCG injection
Phosphate | 72 and 96 hours after hCG injection
cortisol | 72 and 96 hours after hCG injection
total and free testosterone | 72 and 96 hours after hCG injection
total and free estradiol | 72 and 96 hours after hCG injection
albumin, Shbg, VDBP | 72 and 96 hours after hCG injection
25OHD or 24,25OH2D3 | 72 and 96 hours after hCG injection
bone factors such as CTX, osteocalcin, RANKL, FGF23 | 72 and 96 hours after hCG injection
LHCGR | 72 and 96 hours after hCG injection
  in serum
kidney function | 72 and 96 hours after hCG injection
  eGFR/creatinine

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Growth and Reproduction, Rigshospitalet, Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
share all available data through danish data archive
Supporting Information: Study Protocol
Time Frame: 2 years after study completion